CLINICAL TRIAL: NCT06039085
Title: Microendoscopic Electrical Impedance Sensing for Real-time Intraoperative Surgical Margin Assessment
Brief Title: Microendoscopic EI Sensing for Real-time Intraoperative Surgical Margin Assessment
Acronym: RARP EI
Status: Recruiting | Type: Observational
Sponsor: Ryan J. Halter (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Ryan J. Halter, Investigator and Regulatory Sponsor, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: STUDY02001660
Record Dates: First submitted 2023-08-31; First posted 2023-09-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Impedance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: custom device to demonstrate a significant difference in electrical impedance signatures — Custom device will be used to measure electrical impedance signatures.

SUMMARY:
This research will study a custom device developed to detect if any prostate cancer tissue is left behind when the prostate is removed. This device is called an Electrical Impedance Imaging (EII) probe.

DETAILED DESCRIPTION:
Two hundred men will be recruited to participate in this trial. Consent will be obtained from all participating men prior to surgery.

The trial will consist of recording EII data from:

1. In vivo pelvic floor and peri-prostatic tissues remaining after the prostate has been resected
2. Resected ex vivo prostate following extraction from the abdomen (in the OR)
3. Resected ex vivo prostate when transferred to Pathology, post-RARP

The study team will also track post-surgical complications due to the study's technology (e.g., infection) and additional time required to deploy the study technology used to assess feasibility of clinical integration of the EII device. Post-RARP pathological assessment of margin tissues will be used to train and evaluate the study's classification schemes for identifying Positive Surgical Margin (PSMs).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of prostate cancer requiring RARP.
2. Ability to understand and the willingness to sign a written informed consent document.
3. Age ≥ 18 years old

Exclusion Criteria:

1. Adults with implanted electrical devices such as pacemakers
2. Prisoners
3. Adults with impaired decision-making capacity
4. Any condition for which, in the opinion of the investigator, contraindicates study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will be biologically male due to this study's focus on prostate cancer
Study Population: Men with a diagnosis of prostate cancer who require surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Electrical impedance difference between positive and negative surgical margins | 2023-2025
  Outcome measures will include how significantly different electrical impedance signatures are between impedance recordings of positive and negative surgical margins as acquired during prostate surgery.

SECONDARY OUTCOMES:
Safety of EI sensing in vivo electrical sensing | 2023-2025
  Secondary outcome measures will include number of study-related adverse events documented.
Efficacy of EI sensing in vivo electrical sensing | 2023-2025
  Tertiary outcome measures will include classification accuracy of EI-based surgical margin assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Halter, PhD, Principal Investigator — Dartmouth-Hitchcock, Manchester
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No